CLINICAL TRIAL: NCT00093119
Title: A Phase II Trial of ABI-007 in Previously Treated Patients With Metastatic Melanoma
Brief Title: Trial of ABI-007 in Previously Treated Patients With Metastatic Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA014
Record Dates: First submitted 2004-10-01; First posted 2004-10-04 (Estimated); Last update posted 2017-04-26 (Actual); Status verified 2017-04

CONDITIONS: Melanoma; Metastases
Keywords: Metastatic Melanoma
MeSH Terms: conditions — Melanoma; Neoplasm Metastasis | interventions — Albumin-Bound Paclitaxel

INTERVENTIONS:
Drug: ABI-007

SUMMARY:
This trial will treat patients previously treated for advanced (metastatic) melanoma (skin cancer) with a new chemotherapeutic medicine. The new chemotherapy will be administered weekly in cycles of three weekly doses followed by one week rest. A minimum of three cycles of therapy will be given to determine the anti-tumor response of the new chemotherapy. Patients may continue to stay on therapy a maximum of 9-12 cycles if treatment shows continuing benefit.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed Metastatic Melanoma
* At least 18 years old
* No other active malignancy
* Hemoglobin at least 9
* Platelet Count at least 100,000 cells/mm3
* ANC at least 1500 cells/mm3
* AST & ALT less than 2.5X upper limit of normal
* Total bilirubin less than 1.5mg/dL
* Creatine less than 1.5 mg/dL
* Alkaline phosphatase less than 2.5X upper limit of normal
* Life expectancy of at least 12 weeks
* ECOG performance status of 0-1
* Patient must provide informed consent
* Patient must provide authorization to disclose

Exclusion Criteria:

* Evidence of active brain metastases
* The only evidence of metastasis is lytic or blastic bone metastases
* Pre-existing peripheral neuropathy of NCI Toxicity Criteria Scale of grade greater than 2
* Received radiotherapy in last 4wks, except if to a non-target lesion only
* Clinically significant concurrent illness
* Investigator's opinion that patient unlikely to complete study
* Cytotoxic chemotherapeutic agent treatment or investigational drug within previous 4wks
* History of allergy/hypersensitivity to study drug
* Serious Medical Risk Factors determine by the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2003-07; Primary Completion 2005-02 (Actual)

PRIMARY OUTCOMES:
Determine anti-tumor activity of ABI-007 in patients with metastatic melanoma.

SECONDARY OUTCOMES:
Evaluate number of cycles required before patients achieve maximum response

CONTACTS AND LOCATIONS:
Overall Officials: Michael Hawkins, Study Director — Celgene Corporation
Locations (1):
- Abraxis BioScience Inc., Durham, North Carolina, United States